CLINICAL TRIAL: NCT06020625
Title: Mutational Oncology in Clinical Practice: Development of a Comprehensive Cancer Genome Profile Pathway.
Brief Title: Mutational Oncology in Clinical Practice
Acronym: FPG-500
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 3837
Record Dates: First submitted 2023-05-08; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-05

CONDITIONS: Genome Instability; Genetic Predisposition to Disease; Gene Rearrangement
MeSH Terms: conditions — Genomic Instability; Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental)
  Interventions: Genetic: Diagnostic Test

INTERVENTIONS:
Genetic: Diagnostic Test — In order to proceed with molecular characterization, the tumor sample already taken for histological diagnosis will undergo DNA and RNA extraction, which will be analyzed for qualitative and quantitative evaluation. Based on the quantitative data, the method to be used for profiling will be decided.
  Multigenic genomic profiling will be performed for each patient on already taken tumor tissue using different panels depending on the quality and quantity of nucleic acids, in particular the following will be used: comprehensive Genome Profiling (CGP, ≥500 genes), if at least 40 ng of material is available; Profiling with identification of actionable mutations by targeted sequencing with panels of size >50 genes, if <40 ng material available.

SUMMARY:
The study of biological profiling is of fundamental importance in the diagnosis and treatment of many diseases, particularly oncological ones, and for this reason, the integration of molecular characterization into clinical practice becomes essential. NGS allows a high number of samples to be sequenced simultaneously, generating a great deal of genomic information in a short time and at reasonable cost. This information is of fundamental importance for the study of oncogenic drivers and gene alterations that may have a prognostic and/or predictive role in response to new molecularly targeted drugs.

Policlinico A. Gemelli has begun a process of internal reorganization of the research infrastructure following its recognition in 2018 as an Institute of Hospitalization and Treatment with Scientific Character (IRCCS) for its commitment to the disciplines of "Personalized Medicine" and "Innovative Biotechnology." In particular, with regard to genomics, will be equipped with a state-of-the-art technological asset that includes a fully automated process for sample preparation and the highest gene sequencing power available today. This condition makes it possible to perform extensive genomic profiling for large numbers of patients at low cost and in reasonable time.

ELIGIBILITY:
- Patients with neoplasm of the lung, breast, ovary, pancreas, prostate, colorectum, melanoma, GIST, thyroid neoplasm, endometrium, and cholangiocarcinoma:

1. BREAST Locally advanced or metastatic, hormone-responsive, HER2-negative breast neoplasm, progressing after endocrine therapy.
2. LUNG Metastatic disease.
3. OVARY Any stage of nonmucinous, non-borderline epithelial carcinoma of the ovary, fallopian tube, or primary peritoneal carcinoma.
4. PANCREAS Metastatic disease.
5. PROSTATE Metastatic castration-resistant disease.
6. COLORECTUM Metastatic disease.
7. MELANOMA Stage IV or stage III undergoing surgery.
8. GIST Profiling of c-KIT in case of metastatic disease or for patients undergoing surgery and of PDGFRα for all patients with inoperable or metastatic disease.
9. THYROID
10. ENDOMETRIUM
11. CHOLANGIOCARCINOMA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Genome Profiling | 5 years
  Evaluate the impact and efficacy of a 500 cancer genes profiling in an Italian referral centre

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

REFERENCES:
- [Derived] Mastrantoni L, Camarda F, Parrillo C, Persiani F, Trozzi R, Pasciuto T, Manfredelli M, Minucci A, De Paolis E, Capasso I, Iacobelli V, Perri MT, Zannoni GF, Fanfani F, Scambia G, Nero C. Gene actionability according to the ESMO Scale for Clinical Actionability of molecular Targets (ESCAT) in No Specific Molecular Profile (NSMP) endometrial cancer. ESMO Open. 2025 Sep;10(9):105755. doi: 10.1016/j.esmoop.2025.105755. Epub 2025 Sep 3. PMID 40907210
- [Derived] Vita E, Scala A, Vitale A, Mastrantoni L, Evangelista J, D'Auria F, Stefani A, Monaca F, Russo J, Horn G, Troisi P, Cosmai A, Polidori S, Di Salvatore M, De Paolis E, Minucci A, Nero C, Trisolini R, Cancellieri A, Scambia G, Tortora G, Bria E. Network analysis of NRG1 variants of uncertain significance (VUSes) in advanced non-small-cell lung cancer and their prognostic role in EGFR-mutant patients treated with first-line osimertinib. ESMO Open. 2025 Sep;10(9):105556. doi: 10.1016/j.esmoop.2025.105556. Epub 2025 Aug 29. PMID 40885102
- [Derived] Vitale A, Mastrantoni L, Russo J, Giacomini F, Giannarelli D, Duranti S, Vita E, Nero C, D'Argento E, Pasciuto T, Giaco L, Di Salvatore M, Panfili A, Stefani A, Cancellieri A, Lococo F, De Paolis E, Livi V, Daniele G, Trisolini R, Minucci A, Margaritora S, Lorusso D, Normanno N, Scambia G, Tortora G, Bria E. Impact of Comprehensive Genome Profiling on the Management of Advanced Non-Small Cell Lung Cancer: Preliminary Results From the Lung Cancer Cohort of the FPG500 Program. JCO Precis Oncol. 2024 Oct;8:e2400297. doi: 10.1200/PO.24.00297. Epub 2024 Oct 7. PMID 39374480